CLINICAL TRIAL: NCT00400192
Title: Prospective Study of the Kinetics and Mechanisms of Transfusion-associated Microchimerism in Injured Patients
Brief Title: Transfusion-Associated Microchimerism in Individuals Receiving a Blood Transfusion After a Traumatic Injury
Status: Completed | Type: Observational
Sponsor: Vitalant Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1362; R01HL083388 (NIH)
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Chimerism; Blood Transfusion; Wounds and Injuries
Keywords: Microchimerism; Injuries; Leukocytes; Immunologic Techniques
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Individuals who experience a traumatic injury often have a significant amount of blood loss and may require a blood transfusion. In some individuals who receive a blood transfusion, white blood cells from the donor's blood may remain in the body for years, a condition known as microchimerism. This study will examine the reasons why microchimerism occurs in some blood transfusion recipients and not others.

DETAILED DESCRIPTION:
Approximately 20% of individuals who suffer a traumatic injury require a blood transfusion; of these, 10% to 15% experience a condition known as transfusion-associated microchimerism. This occurs when white blood cells, or leukocytes, from the donor's blood persist in the recipient long after the transfusion occurs. The genetically distinct donor cells can remain in the individual for decades, and may account for as many as 4% of the white blood cells in the recipient's body. This suggests that the donor cells are tolerated by the recipient's immune system. The purpose of this study is to examine the specific factors that predispose some blood transfusion recipients to develop microchimerism.

In this study, blood samples will be collected from injured individuals who arrive at the University of California at Davis Medical Center. Individuals who receive a blood transfusion, as well as a control group of individuals who do not receive a transfusion, will be approached to enroll in the study. Individuals who agree to participate will have their blood collected at Days 7, 14, and 28 and Months 3 and 6. Study researchers will analyze the blood for evidence of microchimerism. Participants with microchimerism will undergo additional blood collection at Months 12, 18, 24, 30, and 36. Information will be collected from all participants on health status, injury characteristics, hospital care, blood transfusion details, and blood donor characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for a traumatic injury
* Received at least one unit of transfused red blood cells

Exclusion Criteria:

* Currently incarcerated
* Inadequate decision-making capacity of the participant and no available surrogate decision-maker
* Prior bone marrow or solid organ transplantation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2006-11; Primary Completion 2010-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Prevalence and magnitude of transfusion-associated microchimerism | 1, 2 and 4 weeks, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Busch, MD, PhD, Principal Investigator — Vitalant Research Institute
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Utter GH, Owings JT, Lee TH, Paglieroni TG, Reed WF, Gosselin RC, Holland PV, Busch MP. Blood transfusion is associated with donor leukocyte microchimerism in trauma patients. J Trauma. 2004 Oct;57(4):702-7; discussion 707-8. doi: 10.1097/01.ta.0000140666.15972.37. PMID 15514522
- [Background] Utter GH, Owings JT, Lee TH, Paglieroni TG, Reed WF, Gosselin RC, Holland PV, Busch MP. Microchimerism in transfused trauma patients is associated with diminished donor-specific lymphocyte response. J Trauma. 2005 May;58(5):925-31; discussion 931-2. doi: 10.1097/01.ta.0000162142.72817.5c. PMID 15920405
- [Background] Lee TH, Paglieroni T, Utter GH, Chafets D, Gosselin RC, Reed W, Owings JT, Holland PV, Busch MP. High-level long-term white blood cell microchimerism after transfusion of leukoreduced blood components to patients resuscitated after severe traumatic injury. Transfusion. 2005 Aug;45(8):1280-90. doi: 10.1111/j.1537-2995.2005.00201.x. PMID 16078913